CLINICAL TRIAL: NCT01838278
Title: Effectiveness of Vojta Therapy in Motor Development of Preterm Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad de Murcia (Other)
Collaborators: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Principal Investigator, Julio Perez-Lopez, profesor catedratico, phd, Universidad de Murcia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vojta-2013; 03032/PHCS/05 (Registry Identifier: Fund.Seneca Agencia de Ciencia y Tecnología, Murcia)
Record Dates: First submitted 2013-04-18; First posted 2013-04-24 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Movement Disorders
Keywords: Vojta therapy; Exercise Movement Technique; Early intervention
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vojta physiotherapy Method (Experimental): Children in the experimental group or Vojta group, received two weekly sessions of sensory-motor stimulation and two weekly sessions of Vojta physiotherapy. Sensory motor stimulation and Vojta physiotherapy sessions lasted 50 minutes each. A guidance programme was also given to parents to carry out at home to promote the overall development of the child and teach the necessary Vojta method exercises, these were to be performed four times a day for 20 minutes.
  Interventions: Behavioral: Vojta Physiotherapy Method

INTERVENTIONS:
Behavioral: Vojta Physiotherapy Method — Children in the experimental group or Vojta Group, received two weekly sessions of sensory-motor stimulation and two weekly sessions of Vojta Physiotherapy. Sensory motor stimulation and Vojta physiotherapy sessions lasted 50 minutes each. A guidance programme was also given to parents to carry out at home to promote the overall development of the child and teach the necessary Vojta method exercises, these were to be performed four times a day for 20 minutes.

SUMMARY:
- Justification: Prematurely born children have an increased prevalence of neurodevelopment problems in the first two years. Knowledge regarding the effects of early intervention programs is essential to the follow up of these children and the families.

-Hypothesis: The Vojta Therapy Model showed beneﬁcial effects on motor development outcomes reported by Bayley Sales of Infant Development-Second Edition, in the first 18 months of life on European sample.

DETAILED DESCRIPTION:
Premature children constitute a heterogeneous group regarding gestational age, determinants and causes of their premature birth, illnesses that occur during the neonatal period and the socio-economic status of the family. These constraints could cause an increase in the risk of development in this group of children, as well as motor abnormalities, when compared to the population of infants born at full term.

Cerebral Palsy (CP), for example, is the most common neurological disorder in this group of children. So many studies showed the association between CP and prematurity. They have pointed out that the probability of premature infants having CP is eight times higher compared to full-term infants.

Apart from CP other minor motor abnormalities are also present in the range of consequences for the preterm children.

Therefore, if the increase is considered in children born prematurely who survive, on account of developments in neonatal care, and that the frequency of appearance of motor sequel described in them remains constant, it is of crucial importance from social, economic and health aspects to implement strategies to improve outcomes for these children. In this regard, the development of physiotherapy treatments aimed at preterm infants is essential from a prevention and intervention point of view.

At the Region of Murcia/Spain, when one child is born preterm is directed from the Neonatal Intensive Care Unit (NICU), where there has already been established a protocol for immediate referral among hospitals to early intervention services, where an interdisciplinary team develops an individualized and comprehensive intervention plan according to the characteristics and conditions of each child and, from the motor point of view, the physiotherapist team will be the one who determines the most appropriate action to be taken.

According Vojta, the basic motor function of human has developed in the course of the first year of life, in a process named Postural and Motor Ontogenesis. The practice of Vojta Therapy (VT) had proved to be effective at the treatment of neuromuscular disturbs. Finally, another researches emphasize the importance of follow up of premature children, due to some problems capable of causing motor disability that might not be detectable in the first moments of life, therefore a longitudinal follow-up is recommended.

Regarding this matter, the general aim of this study is to compare the efficiency of the VT on children motor development opposed to other physiotherapy intervention methods used with premature infants without neurological damage, throughout the first 18 months of life, and taking a group of full term infants as a reference. In order to do so, using a longitudinal research design, referring to four different age-groups where children were followed from the first trimester of life until 18 months, corrected age for premature infants and chronologically for full term infants.

- METHODS: This is a longitudinal research design with four assessment follow up during the first trimester (1), at 6, 12 and 18 months. The children are divided into three groups. An experimental group with premature children treated with Vojta Therapy a control group with premature children treated with other traditional physiotherapy methods and another control group (Group 3) with full term infants presenting no risk or pathology.

* Instrument: In order to measure motor development, all children in the experimental group and control groups A and B are evaluated with the Bayley-II scales, in particular with the Psychomotor Scale. The Bayley Scales of Infant and Toddler Development (BSID-II) are a set of standardized rating scales, which enable us to assess the mental, psychomotor and behavioral development of children between 1 and 42 months
* Samples:

The experimental group is composed by preterm children (<37 weeks gestational age), that presented psychomotor delay, but who were not diagnosed with any neurological damage and were receiving VT as a method of physiotherapy treatment, as well as a programme of early intervention including sensory-motor stimulation. This group consists the boys and girls treated at the Early Intervention Centre of Lorca and Aguilas/ Murcia, Spain.

The control group A consists of premature children with similar base characteristics to the experimental group ones who did not receive VT but another method of physiotherapy treatment within a global programme of early intervention that included sensory-motor stimulation. These children are treated and monitored by the Early Intervention Service from the Board of Education of the Region of Murcia (Spain).

The control group B is formed by full term infants, without illnesses or risks. Seventy two boys and girls figured in this group. All children were treated and monitored by the Prevention, Promotion of Early Childhood Development and Early Intervention Service at the University of Murcia (Spain). All parents must sign a consent form authorizing the participation of their children in this project.

- Interventions: Children in the experimental group or Vojta group, receive two weekly sessions of sensory-motor stimulation and two weekly sessions of Vojta Physiotherapy. Sensory motor stimulation and Vojta physiotherapy sessions last 50 minutes each. A guidance programme is also given to parents to carry out at home to promote the overall development of the child and teach the necessary Vojta Method exercises, these are to be performed four times a day for 20 minutes.

Children in control group A or Non-Vojta group, receive two weekly sessions of sensory-motor stimulation and two weekly sessions of physiotherapy with a different methodology to Vojta. Duration of sessions is the same as in the experimental group, of 50 minutes. A guidance programme is also given to parents to carry out at home to promote the overall development of the child and recommendations are provided regarding postural and motor skills that every child needed to ensure proper handling at home.

Children in control group B or the full term infant group receive no intervention of any type but parents are given pointers to promote development at home.

Interventions regarding sensory-motor stimulation in the Early Intervention Centre and guidelines for full term children are carried out by psychologists and specialists in Early Intervention.

Vojta Physiotherapy interventions are performed by expert physiotherapists trained in the method by Vojta Association International.

ANALYSIS OF THE RESULTS All data are analyzed using the computerized statistical package SPSS 15.0 for Windows.

In order to verify our objective, the efficiency of the Vojta Method in motor development of preterm children in the first 18 months of life compared to other physiotherapy methods and using a full term infant group as a reference, mixed 2-factor ANOVA (3x4) with an inter-subject factor (type of sample) with three levels (Vojta, Non-Vojta and Full Term) and one intra-subject factor of repeated assessment (motor development) with 4 measurement times (first trimester, 6, 12 and 18 months) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Experimental Group: First measurement had to be performed during the first trimester of life, from zero to three months corrected age or chronologically depending on the condition of the preterm or full-term infant. Not Diagnosed with any neurological damage and were receiving VT as a method of physiotherapy treatment.
* The A control group: Consisted of premature children with similar base characteristics to the experimental group ones who did not receive VT but another method of physiotherapy treatment within a global programme of early intervention that included sensory-motor stimulation
* The B control group: The control group B was formed by full term infants, without illnesses or risks. Seventy two boys and girls figured in this group. All children were treated and monitored by the Prevention, Promotion of Early Childhood Development and Early Intervention Service at the University of Murcia (Spain).

Exclusion Criteria:

* Experimental, A and B Groups:Parents don't signed a consent form authorizing the participation of their children in this project

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Performance in Psychomotor Subscale - Bayley Scales of Infant and Toddler Development (BSID-II) | 30 days
  Bayley-II scales, in particular with the Psychomotor Scale. The Bayley Scales of Infant and Toddler Development (BSID-II) are a set of standardized rating scales, which enable us to assess the mental, psychomotor and behavioural development of children between 1 and 42 months

SECONDARY OUTCOMES:
Performance Cognitive in Subscale of Bayley-II Scales | 30 days
  Bayley-II scales, in particular with the Cognition Scale. The Bayley Scales of Infant and Toddler Development (BSID-II) are a set of standardized rating scales, which enable us to assess the mental, psychomotor and behavioural development of children between 1 and 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Julio PL Perez-Lopez, Phd, Study Director — Universidad de Murcia; Francisco FR J. Fernández-Rego, MD, Principal Investigator — Universidad de Murcia; María Isabel CG Casbas-Gómez, MD, Study Chair — Early Intervention Centre "Fina Navarro López" of Lorca City Council. Murcia. Spain; María Teresa MF Martínez-Fuentes, Phd, Study Chair — Universidad de Murcia; Angela DH Díaz-Herrero, PHd, Study Chair — Universidad de Murcia; Alfredo BN G. Brito de la Nuez, Phd, Study Chair — Universidad de Murcia; Tatiana Izabele SR Jaworski de Sa Riechi, PHd, Study Chair — Federal University of Parana - Brazil

REFERENCES:
- [Background] Spittle AJ, Anderson PJ, Lee KJ, Ferretti C, Eeles A, Orton J, Boyd RN, Inder T, Doyle LW. Preventive care at home for very preterm infants improves infant and caregiver outcomes at 2 years. Pediatrics. 2010 Jul;126(1):e171-8. doi: 10.1542/peds.2009-3137. Epub 2010 Jun 14. PMID 20547650
- [Background] Kodric J, Sustersic B, Paro-Panjan D. Assessment of general movements and 2.5 year developmental outcomes: pilot results in a diverse preterm group. Eur J Paediatr Neurol. 2010 Mar;14(2):131-7. doi: 10.1016/j.ejpn.2009.04.012. Epub 2009 Jun 21. PMID 19540782
- [Background] Brandt S, Lonstrup HV, Marner T, Rump KJ, Selmar P, Schack LK, d'Avignon M, Noren L, Arman T. Prevention of cerebral palsy in motor risk infants by treatment ad modum Vojta. A controlled study. Acta Paediatr Scand. 1980 May;69(3):283-6. doi: 10.1111/j.1651-2227.1980.tb07079.x. PMID 7376854
- [Background] Yigit S, Kerem M, Livanelioglu A, Oran O, Erdem G, Mutlu A, Turanli G, Tekinalp G, Yurdakok M. Early physiotherapy intervention in premature infants. Turk J Pediatr. 2002 Jul-Sep;44(3):224-9. PMID 12405434
- [Background] Heathcock JC, Lobo M, Galloway JC. Movement training advances the emergence of reaching in infants born at less than 33 weeks of gestational age: a randomized clinical trial. Phys Ther. 2008 Mar;88(3):310-22. doi: 10.2522/ptj.20070145. Epub 2007 Dec 20. PMID 18096650
- [Background] Cameron EC, Maehle V, Reid J. The effects of an early physical therapy intervention for very preterm, very low birth weight infants: a randomized controlled clinical trial. Pediatr Phys Ther. 2005 Summer;17(2):107-19. doi: 10.1097/01.pep.0000163073.50852.58. PMID 16357661
- [Background] McGowan JE, Alderdice FA, Holmes VA, Johnston L. Early childhood development of late-preterm infants: a systematic review. Pediatrics. 2011 Jun;127(6):1111-24. doi: 10.1542/peds.2010-2257. Epub 2011 May 29. PMID 21624885
- [Result] Arnaud C, Daubisse-Marliac L, White-Koning M, Pierrat V, Larroque B, Grandjean H, Alberge C, Marret S, Burguet A, Ancel PY, Supernant K, Kaminski M. Prevalence and associated factors of minor neuromotor dysfunctions at age 5 years in prematurely born children: the EPIPAGE Study. Arch Pediatr Adolesc Med. 2007 Nov;161(11):1053-61. doi: 10.1001/archpedi.161.11.1053. PMID 17984407
- [Result] Evensen KA, Skranes J, Brubakk AM, Vik T. Predictive value of early motor evaluation in preterm very low birth weight and term small for gestational age children. Early Hum Dev. 2009 Aug;85(8):511-8. doi: 10.1016/j.earlhumdev.2009.04.007. Epub 2009 May 17. PMID 19450939
- [Result] Petrini JR, Dias T, McCormick MC, Massolo ML, Green NS, Escobar GJ. Increased risk of adverse neurological development for late preterm infants. J Pediatr. 2009 Feb;154(2):169-76. doi: 10.1016/j.jpeds.2008.08.020. Epub 2008 Dec 10. PMID 19081113